CLINICAL TRIAL: NCT04855123
Title: Evaluation of the Degradation of Renal Function Post Nephrectomy According to Retinal Vascularisation Parameters "NEPHRIN"
Brief Title: Evaluation of the Degradation of Renal Function Post Nephrectomy According to Retinal Vascularisation Parameters
Acronym: NEPHRIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LEGENDRE APJ 2019
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Nephrostomy; Retinal Vascularisation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Other)
  Interventions: Other: retinal imaging; Other: paraclinical surveillance

INTERVENTIONS:
Other: retinal imaging — OCT-angiography, Retinophotography, ocular fundus, Pulsed air tonometer
Other: paraclinical surveillance — blood and urine sampling, assessment of kidney function with creatinine, protein, albumin levels and CKD-EPI equation)

SUMMARY:
Chronic kidney failure in the single remaining kidney is one of the dreaded complications of nephrectomy in patients operated on for cancer-related reasons (1). Indeed, chronic kidney disease (CKD) is associated with major cardiovascular morbidity and mortality (2).

To date, there are few non-invasive methods available to predict the onset and progression of CKD in patients for whom nephrectomy is indicated. Preoperative creatinine and glomerular filtration rate are poor predictors of the subsequent risk of single kidney failure (1). Early predictive markers could help anticipate the management of CKD in patients for whom progression to end-stage renal disease is predictable. Furthermore, such markers could be used as a decision-making aid to specify the type of nephrectomy to be preferred (total versus partial nephrectomy).

The state of microcirculation, particularly retinal, is correlated with the progression of certain conditions such as diabetic nephropathy (3-5). A new technique for evaluating retinal microcirculation called OCT-A (an imaging technique in ophthalmology allowing a precise non-invasive study of the retinal microvascular network) has recently been used by our team to highlight an association between retinal vascularisation and the level of cardiovascular risk in a population of coronary patients without diabetes (6).

We hypothesize that the observation of retinal vascular abnormalities could reflect changes in kidney structure that could underlie chronic renal failure. The aim of this work is thus to evaluate whether the presence of abnormalities in the retinal microvascularisation is 1) predictive of the deterioration in renal function one year after nephrectomy for cancer-related reasons and 2) correlated with renal histological abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Indication for total nephrectomy for kidney cancer decided with a multidisciplinary oncology consultation
* Kidney scan images available
* Patient affiliated to French national health insurance
* Patient who has given oral consent

Exclusion Criteria:

* Pregnant woman
* Ophthalmologic history (macular vascular or degenerative diseases, epiretinal membranes, glaucoma)
* Cannot sit still for 60 minutes
* Metastatic cancer
* Single functional kidney before nephrectomy
* Estimated Glomerular Filtration Flow Rate (CKD-EPI formula) less than 60 mL/min/1.73m2
* Diabetes type 1 or type 2
* Proteinuria at inclusion (or in the 3 months prior to inclusion) on sample with a protein/creatinuria ratio greater than 1g/g or over 24 hours greater than 1g/day
* HIV, HCV or HBV positive serology
* Patient subject to a measure of legal protection (guardianship, curatorship, etc.)

SECONDARY EXCLUSION CRITERIA

* Patient with increased pressure during the measurement of the intraocular pressure before dilation
* Patient with histological abnormalities suggestive of nephropathy (excluding nephroangiosclerosis) or ischemic parenchymal sequelae of renal vein thrombosis in the pathological analysis of the nephrectomy sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Decline in renal function one year after nephrectomy | One year after nephrectomy
  defined in a given patient as the occurrence of a Glomerular Filtration Flow Rate (CKD/EPI equation) of less than 60ml/min/1.73 m2

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France